CLINICAL TRIAL: NCT02834078
Title: Effect of 'Berberine Glucogold' [BGG] on Glucose Metabolism in Individuals With Marginally Impaired Glucose Metabolism Along With Other Markers of Metabolic Syndrome
Brief Title: Effect of BGG on Glucose Metabolism and Other Markers of Metabolic Syndrome
Acronym: Glucogold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Healthy Directions, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD/150301/BGG/PD
Record Dates: First submitted 2016-07-06; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Pre Diabetes
Keywords: HbA1c; Pre Diabetes; Berberine
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BGG (Experimental): Dose: 01 tablet three times daily just before all major meals (breakfast, lunch and dinner)
  Interventions: Dietary Supplement: BGG
- Placebo (Placebo Comparator): Matching placebo capsules [for BGG tablet] composed of micro crystalline cellulose and added colors and odors. Dose: 01 tablet three times daily just before all major meals (breakfast, lunch and dinner)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BGG
  Arms: BGG
Other: Placebo
  Arms: Placebo

SUMMARY:
According to the International Diabetes Federation, one in every 12 individuals is a diabetic (about 8% of the world population). Major risk factors of diabetes are all the aspects of modern life which include obesity, over-weight, high-risk behavior like smoking, alcohol, multiple drug use-recreational or prescribed, environmental risk factors like inactivity and lack of exercise. However there is a window of opportunity between health and disease, which is pre-diabetes.

Pre-diabetes has been defined by American Diabetes Association as Impaired Glucose Tolerance (IGT) which is 7.8 -11.0 mmol/l, Impaired Fasting Glucose Test (IFT) which is 5.6-6.9mmol/l and now added Glycosylated Hemoglobin (HbA1c) of 5.7% to 6.4%.

Though there are plenty of drugs available for significantly impaired glucose metabolism (including oral hypoglycemic agents and insulin), their use in marginally impaired glucose metabolism is questionable due to risk of untoward hypoglycemia.

On the other hand, herbal products like curcumin, as a single ingredient has poor bioavailability problem that restricts its use as standalone treatment. Inulin works as pre-biotic and help to maintain gut microbiota which is considered as precursor for progress of prediabetes to diabetes. However, it does not have any role in primary pathophysiology of impaired glucose metabolism, i.e. pancreatic β cell dysfunction, insulin resistance, hepatic gluconeogenesis or intestinal glucose absorption. Resveratrol and omega-3 basically work on anti-oxidant pathways.

None of these popular ingredients has been studied for their role in structural and functional health of pancreatic β cells which is very important for prediction of further progress of marginally impaired glucose metabolism to significantly impaired glucose metabolism.

It is an unmet need to develop a product which not only improves insulin sensitivity, but also help to preserve the structural and functional health of pancreatic β cells. It also needs to improve overall metabolic and endothelial health of the person considering the close association between impaired glucose metabolism and these parameters.

The proposed supplement - "Berberine GlucoGold "- is an improved version of successfully marketed supplement - Berberine GlucoDefense. It has a balanced composition in which all the ingredients complement each other in such a way that along with the individual role in glucose metabolism it also takes care of overall bioavailability and stability of the supplement. As per the previous data on ingredients, the supplement is also expected to preserve the structural and functional health of pancreatic β cells. The ingredients are also known to have positive effect on overall metabolic and endothelial health. Thus BGG has been developed to address the unmet needs in the area of glucose metabolism and overall metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent.
* Treatment naïve male-female aged 20-60 years of age.
* BMI ≥ 25 kg/m²
* Oral glucose tolerance test (OGTT) ≥140 and ≤250 mg/dl (pre-diabetes and early diagnosed diabetes within 45 days of diagnosis)
* Patient with chronic stable illness can be included ONLY IF he/she is currently NOT on any of the medications included in prohibited list of medicines.
* Currently on herbal supplements can be included after a wash-out period of 7 days.
* Subjects willing to abstain from nicotine and alcohol in the duration of the study.

Exclusion Criteria:

* Subjects with OGTT<140 mg/dl or ≥ 250 mg/dl
* Current treatment with diabetes medications, including metformin
* Current treatment with glucocorticoids
* History of clinically significant hematological, hepatic or renal diseases, as per investigator discretion
* Uncontrolled chronic disease
* Hormonal Disorders
* Subjects on Steroids
* Subjects on Statins
* Chronic inflammatory diseases requiring any medication
* Migraine, Sinusitis
* Subjects Consuming NSAIDS for long term
* Medications include the drugs of prohibited range.
* Pregnant and lactating females.
* Subjects addicted to nicotine, alcohol or any other recreational drug.
* Subjects who are planning to fast for more than 4 days/ per month during the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Oral Disposition Index | Day 0, Day 28, Day 56 and Day 84
Change in Glycated hemoglobin | Day 0, Day 28, Day 56 and Day 84

SECONDARY OUTCOMES:
Change in Fasting blood sugar | Day 0, Day 28, Day 56 and Day 84
Change in Body Mass Index | Day 0, Day 28, Day 56 and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Patil, M.D., Principal Investigator — Maharashtra Council of Indian Medicine; Rajesh Kewalramani, M.B.B.S., Principal Investigator — Maharashtra Council of Indian Medicine

IPD SHARING:
Plan to Share IPD: No